CLINICAL TRIAL: NCT04826042
Title: : Effect of Epidural Injection of Normal Saline or Contrast Medium on Optic Nerve Sheath Diameter
Brief Title: Effect of Contrast Medium on Optic Nerve Sheath Diameter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Ji Hee Hong, professor, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-01-042
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Optic Nerve Sheath Diameter
Keywords: optic nerve sheath diameter

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- contrast group (Active Comparator): injection of contrast medium 6 cc during thoracic epidural catheterization
  Interventions: Other: thoracic epidural catheterization
- normal saline group (Placebo Comparator): injection of normal saline 6 cc during thoracic epidural catheterization
  Interventions: Other: thoracic epidural catheterization

INTERVENTIONS:
Other: thoracic epidural catheterization — thoracic epidural catheterization

SUMMARY:
One method of indirect measurement of intracranial pressure is using optic nerve sheath diameter. There is no study whether equal volume of contrast medium injection has any increasing effect of optic nerve sheath diameter.

This study is designed to measure the changes of optic nerve sheath diameter and cerebral oxygenation when equal volume of contrast medium or normal saline was injected in epidural space.

DETAILED DESCRIPTION:
Previous study showed that different volume of injections (1.0 ml/kg vs. 1.5 ml/kg) during caudal anesthesia showed siginifiant increase of optic nerve sheath diameter in group of high volumes. Increase of ICP can result in harmful effect including reduced cerebral flow and oxygen saturation. Also, increase of ICP can cause headache, syncope and transient loss of visual acuity. The proven and valid method of measuring ICP indirectly is using optic nerve sheath diameter. This study was designed to examine the changes of optic nerve sheath diameter and cerebral oxygenation when equal volume of contrast medium or normal saline was injected in epidural space.

ELIGIBILITY:
Inclusion Criteria:

* lung cancer
* liver cancer
* stomach cancer
* pancreas cancer
* gallbladder

Exclusion Criteria:

* coagulopathy
* infection
* previous spine fusion at thoracic level
* previous brain lesion

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-08-29 (Actual)

PRIMARY OUTCOMES:
optic nerve sheath change during 4 time period | Baseline, 10 minutes, 20 minutes, 40 minutes after the completion of the intervention
  optic nerve sheath change during 4 time period using ultrasound

SECONDARY OUTCOMES:
cerebral oxygenation change during 4 time period | Baseline, 10 minutes, 20 minutes, 40 minutes after the completion of the intervention
  cerebral oxygenation change during 4 time period using cerebral oximeter

CONTACTS AND LOCATIONS:
Locations (1):
- Ji Hee Hong, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hong JH, Park JH, Park KB. Comparison of Increase in the Optic Nerve Sheath Diameter between Epidural Saline and Contrast Medium Injections. Pain Physician. 2022 Mar;25(2):E263-E269. PMID 35322981